CLINICAL TRIAL: NCT06119503
Title: Peer Delivered Episodic Future Thinking to Improve MOUD Treatment Engagement Among Returning Citizens - A Randomized Controlled Trial
Brief Title: Peer-Delivered Episodic Future Thinking for Returning Citizens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Collaborators: Detroit Recovery Project INC (Unknown); Michigan State University (Other); University of Kansas (Other)
Responsible Party: Principal Investigator, Julia Felton, Principal Investigator, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: JRCT: 16686-01
Record Dates: First submitted 2023-10-25; First posted 2023-11-07 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Behavior, Health
Keywords: delay discounting; episodic future thinking; returning citizen; substance use recovery
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Elongating Time HOrizons for Reentry (ETHoR) (Experimental): Episodic Future Thinking (EFT) utilizes participant-generated descriptions of future events to elongate an individual's temporal horizon. In EFT paradigms, the participant is asked to create and envision vivid descriptions of specific, positively valanced, events that could happen in the future. Recent research suggests that directing EFTs to focus on specific goals (i.e. evoking images of oneself engaging in activities consistent with a desired future outcome) are associated with stronger decreases in undesirable health behaviors. Thus, as part of the ETHoR condition, participants will be asked to verbally describe and imagine four specific events reflecting positive activities in which the participant engages in substance and incarceration-free activities, corresponding to predetermined future timepoints. The PRC will encourage participants to include as many contextual and emotional details as possible.
  Interventions: Behavioral: Elongating Time HOrizons for Reentry (ETHoR)
- Standardized Recent Thinking (ERT) (Active Comparator): Individuals in the control group utilizes SET; an approach that controls for activation of episodic thinking but does not engage prospection (the hypothesized mechanism of episodic future thinking, future outcome) are associated with stronger decreases in undesirable health behaviors. Thus, as part of the SET condition, participants will be asked to verbally describe and imagine four current events reflecting positive activities in which the participant engages in substance and incarceration-free activities, corresponding to current experiences. The PRC will encourage participants to include as many contextual and emotional details as possible.
  Interventions: Behavioral: Standardized Episodic Thinking (SET)

INTERVENTIONS:
Behavioral: Elongating Time HOrizons for Reentry (ETHoR) — The adapted episodic future thinking (EFT) intervention will focus on generation of vivid, substance-free, rewarding events that could happen in an incarceration free future.
  Other Names: Episodic Future Thinking (EFT)
  Arms: Elongating Time HOrizons for Reentry (ETHoR)
Behavioral: Standardized Episodic Thinking (SET) — In the standardized episodic thinking (SET) condition, the participant will instead describe in vivid details events that have occurred in the recent past.
  Arms: Standardized Recent Thinking (ERT)

SUMMARY:
The goal of this study is to examine the effectiveness of a brief, episodic future thinking (EFT) intervention in a substance use treatment setting serving returning citizens with substance use disorders (SUD).

The main questions it aims to answer are:

1. Determine preliminary implementation potential of the EFT intervention, including acceptability and feasibility of conducting the intervention.
2. Examine the preliminary effectiveness of this approach, with a specific focus on patient outcomes, including changes in delay discounting, treatment retention, treatment motivation, and substance use.

Participants will be asked to participant in pre and post assessment questionnaires, participate in a single-episode brief intervention followed by tailored phone call follow-ups.

DETAILED DESCRIPTION:
Returning citizens with substance use disorders (SUD) are at the greatest risk for overdose in the first two weeks following the transition from incarceration. Thus, the reentry period is of specific importance for ensuring individuals are engaged and retained in specialized intervention services. Individuals also face numerous, and highly impactful, decisions during this period. They are required to navigate complex tasks (finding employment, securing housing), often with limited financial and social supports. Of particular concern, recent research suggests that the reentry period, often characterized by instability and limited resources, may reinforce a decision-making approach that favors meeting immediate needs relative to engaging in long-term planning. This focus on attaining smaller but immediately available rewards relative to larger, delayed, rewards (known as delay discounting), in turn, has been associated with a number of negative health outcomes, including substance use and poor treatment outcomes (higher dropout and lower motivation). In other words, the reentry context may create an environment which reinforces individuals' tendencies to engage in short-term, reward-seeking behaviors (e.g. substance use, skipping treatment appointments) at a time when their decisions have highly significant consequences (relapse, recidivism). This study will examine the efficacy of implementing a low-cost, brief intervention (Episodic Future Thinking) targeting the reduction of delay discounting with the reentry population to inform broader public health efforts aimed at reducing substance misuse and improvements in treatment outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age
2. Experience in an incarceration setting within 12 months
3. Identify as an individual in substance use recovery
4. Willing to participate in the study
5. Able to participate in written assessments and an intervention conducted in English
6. Willing to receive brief bi-weekly check-in calls for one month, email, and other phone messages related to study participation including SMS/text messages as needed

Exclusion Criteria:

1. Individuals' ineligible or unwilling to participate in study activities and assessments
2. Self-reporting of active and untreated psychosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-11-14 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
Change in Delay Discounting 5 Trial Adjusted Measure | Baseline and up to 3 months post-intervention
  The computer based adjusting amount discounting task uses an adjusting algorithm to determine the amount of immediately available money that is equivalent to a large sum that is delayed by seven discrete durations of time presented in a randomized order (i.e., 1 day, 1 week, 1 month, 6 months, 1 year, 5 years, and 25 years). At each delay, a choice is first presented between the delayed larger sum and a smaller sum available immediately. For each trial, the position of the delayed and immediate amounts are randomly assigned and the participant chooses the preferred option by pressing the corresponding response button.
Change in Consideration of Future Consequences Scale | Baseline and up to 3 months post-intervention
  The Consideration of Future Consequences Scale1 (CFCS-14) is a 14-item self-report questionnaire that assesses active consideration of longer-term implications of an individual's actions. Lower scores on the CFCS-14 are associated with a greater focus on immediate needs and have been found to be associated with less engagement in health behaviors1819 and greater substance use. The measure has been used extensively among adult samples and demonstrates strong reliability and validity. Research suggests modest but significant correlations with the MCQ.

SECONDARY OUTCOMES:
Change in Short Michigan Alcohol Screening Test (SMAST) | Baseline and up to 3 months post-intervention
  The SMAST is a brief questionnaire consisting of 13 items. It can be completed in just a few minutes and is designed for individuals with a reading level equivalent to that of a 7th grader. This assessment tool was derived from the Michigan Alcoholism Screening Test and has been found to be a reliable diagnostic tool to detect at-risk alcohol use, alcohol abuse, or alcoholism. The evaluation data suggests its effectiveness, with no notable occurrence of false positives.
Change in Drug Abuse Screen Test (DAST) | Baseline and up to 3 months post-intervention
  The DAST offer a concise self-report tool for screening populations, identifying clinical cases, and researching treatment effectiveness related to drug abuse. It is applicable for use with both adults and older adolescents. The DAST-10 provides a numerical gauge of the extent of drug abuse-related consequences. Administering the assessment takes around 5 minutes Condensed from its longer counterpart of 28 items, the DAST-10 comprises 10 self-report items.

CONTACTS AND LOCATIONS:
Locations (1):
- Detroit Recovery Project, Detroit, Michigan, United States

REFERENCES:
- [Background] Zeng S, Minton TD. Jail Inmates in 2019. Bureau of Justice Statistics. Accessed July 15, 2022. https://bjs.ojp.gov/library/publications/jail-inmates-2019
- [Background] Loeffler CE, Nagin DS. The Impact of Incarceration on Recidivism. Annu Rev Criminol. 2022;5(1):133-152. doi:10.1146/annurev-criminol-030920-112506
- [Background] NIDA. Criminal Justice DrugFacts. National Institute on Drug Abuse. Published June 1, 2020. Accessed July 11, 2022. https://nida.nih.gov/publications/drugfacts/criminal-justice
- [Background] Binswanger IA, Blatchford PJ, Mueller SR, Stern MF. Mortality after prison release: opioid overdose and other causes of death, risk factors, and time trends from 1999 to 2009. Ann Intern Med. 2013 Nov 5;159(9):592-600. doi: 10.7326/0003-4819-159-9-201311050-00005. PMID 24189594
- [Background] Pizzicato LN, Drake R, Domer-Shank R, Johnson CC, Viner KM. Beyond the walls: Risk factors for overdose mortality following release from the Philadelphia Department of Prisons. Drug Alcohol Depend. 2018 Aug 1;189:108-115. doi: 10.1016/j.drugalcdep.2018.04.034. Epub 2018 Jun 5. PMID 29908410
- [Background] Garland B, Wodahl EJ, Mayfield J. Prisoner Reentry in a Small Metropolitan Community: Obstacles and Policy Recommendations. Criminal Justice Policy Review. 2011;22(1):90-110. doi:10.1177/0887403409359804
- [Background] Jonson CL, Cullen FT. Prisoner reentry programs. Crime and justice. 2015;44(1):517-575.
- [Background] Solomon AL. From prison to work: The employment dimensions of prisoner reentry. Published online 2004.
- [Background] Hattery AJ, Smith E. Prisoner Reentry and Social Capital: The Long Road to Reintegration. Lexington Books; 2010.
- [Background] Grieb SM, Crawford A, Fields J, Smith H, Harris R, Matson P. "The stress will kill you": prisoner reentry as experienced by family members and the urgent need for support services. J Health Care Poor Underserved. 2014 Aug;25(3):1183-200. doi: 10.1353/hpu.2014.0118. PMID 25130233
- [Background] Amso D, Lynn A. Distinctive Mechanisms of Adversity and Socioeconomic Inequality in Child Development: A Review and Recommendations for Evidence-Based Policy. Policy Insights Behav Brain Sci. 2017;4(2):139-146. doi: 10.1177/2372732217721933. Epub 2017 Jul 25. PMID 30345346
- [Background] Sheridan MA, Peverill M, Finn AS, McLaughlin KA. Dimensions of childhood adversity have distinct associations with neural systems underlying executive functioning. Dev Psychopathol. 2017 Dec;29(5):1777-1794. doi: 10.1017/S0954579417001390. PMID 29162183
- [Background] Wesarg C, Akker ALVD, Oei NYL, Hoeve M, Wiers RW. Identifying pathways from early adversity to psychopathology: A review on dysregulated HPA axis functioning and impaired self-regulation in early childhood. European Journal of Developmental Psychology. 2020;17(6):808-827. doi:10.1080/17405629.2020.1748594
- [Background] Friedel E, Schlagenhauf F, Beck A, Dolan RJ, Huys QJ, Rapp MA, Heinz A. The effects of life stress and neural learning signals on fluid intelligence. Eur Arch Psychiatry Clin Neurosci. 2015 Feb;265(1):35-43. doi: 10.1007/s00406-014-0519-3. Epub 2014 Aug 21. PMID 25142177
- [Background] Mani A, Mullainathan S, Shafir E, Zhao J. Poverty impedes cognitive function. Science. 2013 Aug 30;341(6149):976-80. doi: 10.1126/science.1238041. PMID 23990553
- [Background] Platt JM, McLaughlin KA, Luedtke AR, Ahern J, Kaufman AS, Keyes KM. Targeted Estimation of the Relationship Between Childhood Adversity and Fluid Intelligence in a US Population Sample of Adolescents. Am J Epidemiol. 2018 Jul 1;187(7):1456-1466. doi: 10.1093/aje/kwy006. PMID 29982374
- [Background] Acheson A, Vincent AS, Cohoon A, Lovallo WR. Early life adversity and increased delay discounting: Findings from the Family Health Patterns project. Exp Clin Psychopharmacol. 2019 Apr;27(2):153-159. doi: 10.1037/pha0000241. Epub 2018 Dec 17. PMID 30556730
- [Background] Martinez JL, Hasty C, Morabito D, Maranges HM, Schmidt NB, Maner JK. Perceptions of childhood unpredictability, delay discounting, risk-taking, and adult externalizing behaviors: A life-history approach. Dev Psychopathol. 2022 May;34(2):705-717. doi: 10.1017/S0954579421001607. Epub 2022 Jan 18. PMID 35039110
- [Background] Amlung M, Vedelago L, Acker J, Balodis I, MacKillop J. Steep delay discounting and addictive behavior: a meta-analysis of continuous associations. Addiction. 2017 Jan;112(1):51-62. doi: 10.1111/add.13535. Epub 2016 Sep 1. PMID 27450931
- [Background] Felton JW, Collado A, Ingram K, Lejuez CW, Yi R. Changes in delay discounting, substance use, and weight status across adolescence. Health Psychol. 2020 May;39(5):413-420. doi: 10.1037/hea0000833. Epub 2020 Jan 9. PMID 31916829
- [Background] Audrain-McGovern J, Rodriguez D, Epstein LH, Cuevas J, Rodgers K, Wileyto EP. Does delay discounting play an etiological role in smoking or is it a consequence of smoking? Drug Alcohol Depend. 2009 Aug 1;103(3):99-106. doi: 10.1016/j.drugalcdep.2008.12.019. Epub 2009 May 14. PMID 19443136
- [Background] Stevens L, Verdejo-Garcia A, Roeyers H, Goudriaan AE, Vanderplasschen W. Delay discounting, treatment motivation and treatment retention among substance-dependent individuals attending an in inpatient detoxification program. J Subst Abuse Treat. 2015 Feb;49:58-64. doi: 10.1016/j.jsat.2014.08.007. Epub 2014 Sep 1. PMID 25245429
- [Background] Washio Y, Higgins ST, Heil SH, McKerchar TL, Badger GJ, Skelly JM, Dantona RL. Delay discounting is associated with treatment response among cocaine-dependent outpatients. Exp Clin Psychopharmacol. 2011 Jun;19(3):243-8. doi: 10.1037/a0023617. PMID 21517195
- [Background] Sheffer CE, Christensen DR, Landes R, Carter LP, Jackson L, Bickel WK. Delay discounting rates: a strong prognostic indicator of smoking relapse. Addict Behav. 2014 Nov;39(11):1682-1689. doi: 10.1016/j.addbeh.2014.04.019. Epub 2014 May 5. PMID 24878037
- [Background] Duffy KA, McLaughlin KA, Green PA. Early life adversity and health-risk behaviors: proposed psychological and neural mechanisms. Ann N Y Acad Sci. 2018 Sep;1428(1):151-169. doi: 10.1111/nyas.13928. Epub 2018 Jul 16. PMID 30011075
- [Background] Kim-Spoon J, Lauharatanahirun N, Peviani K, Brieant A, Deater-Deckard K, Bickel WK, King-Casas B. Longitudinal pathways linking family risk, neural risk processing, delay discounting, and adolescent substance use. J Child Psychol Psychiatry. 2019 Jun;60(6):655-664. doi: 10.1111/jcpp.13015. Epub 2019 Feb 27. PMID 30809804
- [Background] Levitt EE, Amlung MT, Gonzalez A, Oshri A, MacKillop J. Consistent evidence of indirect effects of impulsive delay discounting and negative urgency between childhood adversity and adult substance use in two samples. Psychopharmacology (Berl). 2021 Jul;238(7):2011-2020. doi: 10.1007/s00213-021-05827-6. Epub 2021 Mar 29. PMID 33782722
- [Background] Trommsdorff G, Lamm H. Future orientation of institutionalized and noninstitutionalized delinquents and nondelinquents. European Journal of Social Psychology. 1980;10(3):247-278.
- [Background] Arantes J, Berg ME, Lawlor D, Grace RC. Offenders have higher delay-discounting rates than non-offenders after controlling for differences in drug and alcohol abuse. Legal and Criminological Psychology. 2013;18(2):240-253. doi:10.1111/j.2044-8333.2012.02052.x
- [Background] Felton JW, Collado A, Ingram KM, Doran K, Yi R. Improvement of Working Memory is a Mechanism for Reductions in Delay Discounting Among Mid-Age Individuals in an Urban Medically Underserved Area. Ann Behav Med. 2019 Oct 7;53(11):988-998. doi: 10.1093/abm/kaz010. PMID 30955043
- [Background] Chiou WB, Wu WH. Episodic Future Thinking Involving the Nonsmoking Self Can Induce Lower Discounting and Cigarette Consumption. J Stud Alcohol Drugs. 2017 Jan;78(1):106-112. doi: 10.15288/jsad.2017.78.106. PMID 27936370
- [Background] Stein JS, Wilson AG, Koffarnus MN, Daniel TO, Epstein LH, Bickel WK. Unstuck in time: episodic future thinking reduces delay discounting and cigarette smoking. Psychopharmacology (Berl). 2016 Oct;233(21-22):3771-3778. doi: 10.1007/s00213-016-4410-y. Epub 2016 Aug 23. PMID 27553824
- [Background] Snider SE, LaConte SM, Bickel WK. Episodic Future Thinking: Expansion of the Temporal Window in Individuals with Alcohol Dependence. Alcohol Clin Exp Res. 2016 Jul;40(7):1558-66. doi: 10.1111/acer.13112. Epub 2016 Jun 1. PMID 27246691
- [Background] Garcia-Perez A, Aonso-Diego G, Weidberg S, Secades-Villa R. Effects of episodic future thinking on reinforcement pathology during smoking cessation treatment among individuals with substance use disorders. Psychopharmacology (Berl). 2022 Feb;239(2):631-642. doi: 10.1007/s00213-021-06057-6. Epub 2022 Jan 12. PMID 35020047
- [Background] Sze YY, Stein JS, Bickel WK, Paluch RA, Epstein LH. Bleak Present, Bright Future: Online Episodic Future Thinking, Scarcity, Delay Discounting, and Food Demand. Clin Psychol Sci. 2017 Jul;5(4):683-697. doi: 10.1177/2167702617696511. Epub 2017 May 2. PMID 28966885
- [Background] Sze YY, Daniel TO, Kilanowski CK, Collins RL, Epstein LH. Web-Based and Mobile Delivery of an Episodic Future Thinking Intervention for Overweight and Obese Families: A Feasibility Study. JMIR Mhealth Uhealth. 2015 Dec 16;3(4):e97. doi: 10.2196/mhealth.4603. PMID 26678959
- [Background] O'Neill J, Daniel TO, Epstein LH. Episodic future thinking reduces eating in a food court. Eat Behav. 2016 Jan;20:9-13. doi: 10.1016/j.eatbeh.2015.10.002. Epub 2015 Oct 28. PMID 26562686
- [Background] Kaplan BA, Reed DD, Jarmolowicz DP. Effects of episodic future thinking on discounting: Personalized age-progressed pictures improve risky long-term health decisions. J Appl Behav Anal. 2016 Mar;49(1):148-69. doi: 10.1002/jaba.277. Epub 2015 Dec 17. PMID 26679531
- [Background] Dassen FCM, Jansen A, Nederkoorn C, Houben K. Focus on the future: Episodic future thinking reduces discount rate and snacking. Appetite. 2016 Jan 1;96:327-332. doi: 10.1016/j.appet.2015.09.032. Epub 2015 Sep 30. PMID 26431684
- [Background] Rosch SA, Stramaccia DF, Benoit RG. Promoting farsighted decisions via episodic future thinking: A meta-analysis. J Exp Psychol Gen. 2022 Jul;151(7):1606-1635. doi: 10.1037/xge0001148. Epub 2021 Nov 29. PMID 34843367
- [Background] Patel H, Amlung M. Acute and extended exposure to episodic future thinking in a treatment seeking addiction sample: A pilot study. J Subst Abuse Treat. 2020 Sep;116:108046. doi: 10.1016/j.jsat.2020.108046. Epub 2020 Jun 1. PMID 32741499
- [Background] O'Donnell S, Oluyomi Daniel T, Epstein LH. Does goal relevant episodic future thinking amplify the effect on delay discounting? Conscious Cogn. 2017 May;51:10-16. doi: 10.1016/j.concog.2017.02.014. Epub 2017 Mar 8. PMID 28282631
- [Background] Liu L, Feng T, Chen J, Li H. The value of emotion: how does episodic prospection modulate delay discounting? PLoS One. 2013 Nov 28;8(11):e81717. doi: 10.1371/journal.pone.0081717. eCollection 2013. PMID 24312341
- [Background] Van Ginneken E. The role of hope in preparation for release from prison. Prison Service Journal. 2015;220(1):10-15.
- [Background] Vuk M, Applegate BK. From Future Orientation to Readiness for Reentry: An Exploratory Study of Prelease Cognitions of Incarcerated Men. Incarceration. 2021;2(3):26326663211052280. doi:10.1177/26326663211052282
- [Background] Eddie D, Hoffman L, Vilsaint C, Abry A, Bergman B, Hoeppner B, Weinstein C, Kelly JF. Lived Experience in New Models of Care for Substance Use Disorder: A Systematic Review of Peer Recovery Support Services and Recovery Coaching. Front Psychol. 2019 Jun 13;10:1052. doi: 10.3389/fpsyg.2019.01052. eCollection 2019. PMID 31263434
- [Background] Gagne CA, Finch WL, Myrick KJ, Davis LM. Peer Workers in the Behavioral and Integrated Health Workforce: Opportunities and Future Directions. Am J Prev Med. 2018 Jun;54(6 Suppl 3):S258-S266. doi: 10.1016/j.amepre.2018.03.010. PMID 29779550
- [Background] Reif S, Braude L, Lyman DR, Dougherty RH, Daniels AS, Ghose SS, Salim O, Delphin-Rittmon ME. Peer recovery support for individuals with substance use disorders: assessing the evidence. Psychiatr Serv. 2014 Jul;65(7):853-61. doi: 10.1176/appi.ps.201400047. PMID 24838535
- [Background] Victor G, Sightes E, Watson DP, Ray B, Bailey K, Robision L, Fears G, Edwards R, Salyers M. Designing and implementing an intervention for returning citizens living with substance use disorder: discovering the benefits of peer recovery coach involvement in pilot clinical trial decision-making. J Offender Rehabil. 2021;60(2):138-158. doi: 10.1080/10509674.2020.1863301. Epub 2021 Jan 11. PMID 33551628
- [Background] O'Mara-Eves A, Brunton G, McDaid D, Oliver S, Kavanagh J, Jamal F, Matosevic T, Harden A, Thomas J. Community engagement to reduce inequalities in health: a systematic review, meta-analysis and economic analysis. Southampton (UK): NIHR Journals Library; 2013 Nov. Available from http://www.ncbi.nlm.nih.gov/books/NBK262817/ PMID 25642563
- [Background] Brown E, Males M. Does age or poverty level best predict criminal arrest and homicide rates? A preliminary investigation. Justice Policy Journal. 2011;8(1):1-30.
- [Background] Kleinman MB, Felton JW, Johnson A, Magidson JF. "I have to be around people that are doing what I'm doing": The importance of expanding the peer recovery coach role in treatment of opioid use disorder in the face of COVID-19 health disparities. J Subst Abuse Treat. 2021 Mar;122:108182. doi: 10.1016/j.jsat.2020.108182. Epub 2020 Oct 21. PMID 33160763
- [Background] Moore KE, Siebert S, Brown G, Felton J, Johnson JE. Stressful life events among incarcerated women and men: Association with depression, loneliness, hopelessness, and suicidality. Health Justice. 2021 Aug 24;9(1):22. doi: 10.1186/s40352-021-00140-y. PMID 34427798
- [Background] Felton JW, Hailemariam M, Richie F, Reddy MK, Edukere S, Zlotnick C, Johnson JE. Preliminary efficacy and mediators of interpersonal psychotherapy for reducing posttraumatic stress symptoms in an incarcerated population. Psychother Res. 2020 Feb;30(2):239-250. doi: 10.1080/10503307.2019.1587192. Epub 2019 Mar 11. PMID 30857489
- [Background] Stoddard SA, Montgomery BW, Maschino LD, et al. Establishing the Effectiveness of Enhanced Implementation Methods in Preventative Behavioral Health. medRxiv. Published online 2020.
- [Background] Hailemariam M, Felton JW, Key K, Greer D, Jefferson BL, Muhammad J, Miller R, Richie F, Robinson D, Saddler S, Spencer B, Summers M, White JMC, Johnson JE. Intersectionality, special populations, needs and suggestions: the Flint Women's study. Int J Equity Health. 2020 Jan 31;19(1):18. doi: 10.1186/s12939-020-1133-9. PMID 32005120
- [Background] Collado A, Felton JW, Taylor H, Eure A, Yi R. Conscientiousness explains the link between childhood neglect and cigarette smoking in adults from a low-income, urban area-the differential effects of sex. Child Abuse Negl. 2019 Feb;88:152-158. doi: 10.1016/j.chiabu.2018.10.015. Epub 2018 Nov 30. PMID 30508683
- [Background] Collado A, Felton JW, Taylor H, Doran K, Yi R. The Indirect Effects of Trait Anxiety on Drug Use Via Emotion Dysregulation in a Low-Income Sample. Subst Use Misuse. 2020;55(8):1320-1326. doi: 10.1080/10826084.2020.1741631. Epub 2020 Mar 18. PMID 32186420
- [Background] DePietro A. U.S. Poverty Rate By City In 2021. Forbes. Accessed August 15, 2022. https://www.forbes.com/sites/andrewdepietro/2021/11/26/us-poverty-rate-by-city-in-2021/
- [Background] U.S. Census Bureau QuickFacts: Detroit city, Michigan; Michigan. Accessed July 15, 2022. https://www.census.gov/quickfacts/fact/table/detroitcitymichigan,MI/PST045221
- [Background] Weisz JR, Jensen AL, McLeod BD. Development and Dissemination of Child and Adolescent Psychotherapies: Milestones, Methods, and a New Deployment-Focused Model. In: Psychosocial Treatments for Child and Adolescent Disorders: Empirically Based Strategies for Clinical Practice, 2nd Ed. American Psychological Association; 2005:9-39.
- [Background] Daniel TO, Said M, Stanton CM, Epstein LH. Episodic future thinking reduces delay discounting and energy intake in children. Eat Behav. 2015 Aug;18:20-4. doi: 10.1016/j.eatbeh.2015.03.006. Epub 2015 Mar 28. PMID 25863227
- [Background] Proctor E, Silmere H, Raghavan R, Hovmand P, Aarons G, Bunger A, Griffey R, Hensley M. Outcomes for implementation research: conceptual distinctions, measurement challenges, and research agenda. Adm Policy Ment Health. 2011 Mar;38(2):65-76. doi: 10.1007/s10488-010-0319-7. PMID 20957426
- [Background] Miller WR, Tonigan JS. Stages of Change Readiness and Treatment Eagerness Scale (SOCRATES). APA PsycTests. Published online 1996. Accessed September 29, 2021. https://doi.apa.org/doiLanding?doi=10.1037%2Ft00536-000
- [Background] Holt DD, Green L, Myerson J. Is discounting impulsive?. Evidence from temporal and probability discounting in gambling and non-gambling college students. Behav Processes. 2003 Oct 31;64(3):355-367. doi: 10.1016/s0376-6357(03)00141-4. PMID 14580704
- [Background] Satinsky EN, Doran K, Felton JW, Kleinman M, Dean D, Magidson JF. Adapting a peer recovery coach-delivered behavioral activation intervention for problematic substance use in a medically underserved community in Baltimore City. PLoS One. 2020 Jan 31;15(1):e0228084. doi: 10.1371/journal.pone.0228084. eCollection 2020. PMID 32004328
- [Background] Middlemass KM, Smiley C. Prisoner Reentry in the 21st Century: Critical Perspectives of Returning Home. Routledge; 2019.
- [Background] Crapanzano KA, Hammarlund R, Ahmad B, Hunsinger N, Kullar R. The association between perceived stigma and substance use disorder treatment outcomes: a review. Subst Abuse Rehabil. 2018 Dec 27;10:1-12. doi: 10.2147/SAR.S183252. eCollection 2019. PMID 30643480